CLINICAL TRIAL: NCT06972381
Title: Piloting a Patient Navigator Program to Facilitate Uptake and Persistence With Evidence-based Weight Loss Interventions
Brief Title: Piloting a Patient Navigator Program for Weight Loss
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Meghan Butryn, Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DK140184 (NIH)
Record Dates: First submitted 2025-05-01; First posted 2025-05-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
Keywords: weight loss; overweight; obesity; patient navigator; weight loss counselor
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized controlled pilot trial. Participants will be assigned to either the navigator condition or usual care, with a 1:1 allocation
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigator Intervention (Experimental): Participants assigned to the navigator condition will receive a weight loss counselor who they will maintain contact with over the 12 month period. Participants will attend 5-8 videoconferencing sessions with their navigator, as well as communicate with them monthly via email for extra support. Navigators will help participants initiate and adhere to an evidence-based weight loss intervention, without providing the treatment themselves.
  Interventions: Behavioral: Navigator
- Usual Care (No Intervention): Participants assigned to the usual care condition will have no intervention contact during the 12-month data collection period and are encouraged to use resources available to them in community and in their health care system to identify treatment options. They will be given the option to attend a two-hour educational workshop (on videoconferencing software) after the 12-month assessment, to learn more about evidence-based approaches to weight loss.

INTERVENTIONS:
Behavioral: Navigator — Participants in the navigator condition will meet with their counselor for sessions twice in month 1, once in month 2, once in month 4, and once in month 8. Three additional sessions may scheduled if desired by the participant. Navigators will assess treatment preferences, provide information about evidence-based treatment options for weight loss, aid in decision making, and facilitate action during the intervention initiation process. Following initiation of a weight loss treatment, navigators will also assess adherence to and acceptability of the selected weight loss intervention, and engage in problem solving and motivational enhancement to facilitate persistence with the original intervention or provide the support necessary for switching to an alternative intervention option. Additional intervention contact will include monthly emails over the 12 month period. Navigators will receive resource guides to help them tailor sessions to the individual participant.
  Other Names: Weight loss counselor
  Arms: Navigator Intervention

SUMMARY:
Evidence-based interventions for overweight and obesity are underutilized. The utilization and efficacy of these interventions may improve with the implementation of a patient navigator program, as has been practiced in other fields (e.g., cancer). The proposed study will enroll adults ("index participants") (N=68) with overweight/obesity in a 12-month program in which they will be provided with a navigator who will help them understand their options for evidence-based weight loss intervention and who will promote initiation and continued engagement with an intervention option. The project will provide information about how well received the navigator program is and the extent to which it works as expected.

DETAILED DESCRIPTION:
Most adults who attempt weight loss do not use evidence-based interventions; instead, they engage in self-directed dieting, which is typically short-lived and has poor efficacy. These individuals often a) feel overwhelmed by navigating other options in the challenging climate of the U.S. healthcare system, b) lack knowledge about the costs, availability, efficacy and features of various interventions, and c) feel ambivalent about committing to a more structured weight loss approach. This pilot clinical trial is designed to test the use of a weight loss navigation program to address these problems.

In the proposed study, participants (N = 68) will be adults with a BMI > 27 kg/m2, recruited from the community, who are interested in weight loss. Participants will be randomized to either the navigator program or usual care. Usual care will have no intervention contact. Participants in the navigator condition will have 12 months of contact with their assigned counselor. Participants will be asked to attend a minimum of 5 sessions with the counselor conducted via videoconferencing software: two sessions in Month 1, one in Month 2, one in Month 4, and one in Month 8. Three additional sessions can be held at any time if the counselor and participant agree the additional contact would be helpful. Participants and navigators will also maintain contact via email outside of sessions. The navigator's goal will be to connect the participant with another provider or program who can directly deliver a form of evidence-based treatment to the participant (i.e., select commercial programs, behavioral weight loss, counseling from a licensed clinician, prescription medications and bariatric surgery), but the navigator will not be attempting to deliver any of those five evidence-based interventions themself. Navigators will assess treatment preferences, provide information about evidence-based treatment options for weight loss, aid in decision making, and facilitate action during the intervention initiation process.

Outcomes will be measured at months 0, 6, and 12 months. The primary aim is determining if weight loss is higher in the navigator condition. Secondary aims include assessing the feasibility and acceptability of this pilot study and gathering feedback to improve the navigator program for future research. The current study will be a major contribution to the literature, as no evidence is available yet to understand the utility of a navigator program for treatment of overweight and obesity. This program has the potential to make a major public health impact by connecting many more of the millions of adults who could benefit from weight loss intervention with currently available, evidence-based tools.

ELIGIBILITY:
Inclusion criteria include:

* BMI > 27 kg/m2
* weight < 396 pounds due to limits of the wireless scale
* age 18 to 75
* ability to read and speak English sufficiently to engage with a counselor and complete study measures
* willing to be randomized to either study condition
* willing to engage with a counselor for assistance in identifying and initiating a weight loss intervention
* successfully complete enrollment and assessments tasks, including connecting a wireless scale for baseline measurement of weight
* reliable access to a device capable of using email and Drexel approved videoconferencing software
* residing in the greater Philadelphia metropolitan area, which includes Southeastern PA, Southern NJ, Northeast MD, and Northern DE
* agree that they will not join another intervention study in the WELL Center in the next 12 months

Exclusion criteria include:

* a medical or psychiatric condition that may a) limit appropriateness of weight loss intervention or b) be likely to cause a change in weight in the next 12 months (e.g., anorexia nervosa, bulimia nervosa, end-stage kidney disease, some types of cancer)
* currently taking weight loss medication or engaging in any other form of weight management intervention
* history of bariatric surgery
* a calculated weight suppression value of 10% or higher
* currently pregnant or planning to become pregnant in the next 12 months
* adults unable to consent, children, pregnant women, and prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | 0 month, 6 month, 12 month
  Participants will be instructed to use a Withings wireless scale (stated accuracy to 0.1 kg) to weigh themselves. Participants will be instructed to step on the scale in the morning (before eating but after using the bathroom), wearing no shoes and minimal clothing, with the scale on a hard, flat, surface. Participants will be instructed to measure their weight for three consecutive days so that a participant's mean can be calculated at each time point in order to minimize the influence of daily fluctuations of weight. Data will be pulled from the Withings cloud to the study database via the Withings API. In order to maximize accuracy, we will remove errant weights (e.g., >1 kg change in 1 day).

SECONDARY OUTCOMES:
5% weight change | 0, 6, 12 months
  The proportion of participants who have >5% weight loss (which is a standard threshold for clinical significance) will be a secondary outcome.
Recruitment feasibility | Throughout the 7 month recruitment and enrollment period
  Data on recruitment rate will be available via REDCap. The benchmark is to enroll ~10 participants per month over the course of the 7-month recruitment period.
Retention feasibility | 6, 12 months
  Data on retention will be available via REDCap. The benchmark is to retain a minimum of 75% of participants at 6 and 12 months.
Intervention Acceptability | 6 month, 12 month
  Participants in the Navigator condition will be administered the Treatment Acceptability Questionnaire at 6 and 12 months, with content modified as needed to be clear that the items are referring to the navigator program, not any other weight loss intervention the participant may be receiving. This measure has six items, each rated on a 1-7 scale, with 7 being most positive. The benchmark of mean score of 5 or greater in the navigator condition was chosen based on face validity to correspond to ratings that are positive, as opposed to negative or neutral.
Intervention engagement | 0-12 months
  Attendance will be recorded in REDCap, so that the proportion of participants attending 4 or more sessions can be calculated (benchmark = 75%).
Intervention fidelity | 0-12 months
  To assess the feasibility of navigators having fidelity to their assigned intervention approaches, a structured rubric will be created to code 10% of audio- or videorecorded sessions and 10% of emails. Sessions and emails will be randomly selected for review. The rubric will outline ratings for adhering to principles of the intervention approach as well as ratings for contamination. Each item in the rubric will be rated on a 1-10 scale, with 10 showing perfect fidelity. The benchmark of mean score of 8 or higher was chosen based on face validity.
Utilization of Weight Change Interventions | 6 month, 12 month
  A structured interview, conducted by a blinded member of the research staff, will query which types of weight change interventions have been utilized in the previous 6 months, as well as the length of intervention engagement. De-identified data will be coded. Each intervention reported by a participant will be categorized as a specific type of evidence-based intervention (nutritional counseling, behavioral counseling, select commercial programs, pharmacotherapy, or bariatric surgery) or a type of non-evidence-based intervention (e.g., self-guided weight loss attempt, use of herbal supplements, etc.). A categorical variable will capture whether or not the participant received an evidence-based intervention in the previous 6 months. A continuous measure also will indicate the number of weeks in the previous 6 months in which the the participant reported active use of an evidence-based intervention.
Qualitative Feedback | 6 month, 12 month
  Semi-structured interviews (30 minutes each) will be conducted by trained team members at months 6 and 12 to inform improvements in the navigator program for future research. These qualitative data will be collected from 10 program participants in the Navigator condition. Participants will be purposively sampled across personal characteristics (e.g., age, gender), process (adherence, satisfaction), and outcome metrics (utilization of weight loss interventions, weight) to ensure diverse perspectives and insights. Interviews will explore a) acceptability of research and intervention procedures, and b) factors that hinder or facilitate adherence and weight loss.

OTHER OUTCOMES:
Participant characteristics | 0 month
  Self-report information will be collected regarding age, race, ethnicity, sex, gender, income, education, insurance status, employment status, and marital status. These variables will be used for exploratory analyses.
Weight change history | 0 months
  All participants will complete a weight change history questionnaire developed by Myers et al. (2013) at BL.
Comorbidities Checklist | 0 month
  A self-report checklist will ask if the participant has any of the following weight-related comorbidities: hypertension, type 2 diabetes or pre-diabetes, gastroesophageal reflux disease, arthritis, obstructive sleep apnea, heart disease including coronary artery disease or atrial fibrillation or heart failure, dyslipidemia (e.g., high cholesterol), non-alcoholic liver disease.
Attitudes toward weight change treatments | 0 months
  A series of questions developed by the study team will be administered to participants at BL only. These questions assess participant views regarding various evidence-based weight change treatments, and will ask participant to rank these treatments based on their long-term efficacy, accessibility, and trustworthiness with a ranking of 1 being the best, and a ranking of 6 being the worst.
Interest in evidence-based weight loss options | 0 months
  A series of questions developed by Wharton et al. (2016) will be administered to all participants in the form of an online questionnaire at BL only. These questions will assess participant views and level of interest in evidence-based weight loss options i.e., bariatric surgery, anti-obesity medications, behavioral weight loss interventions, nutrition counseling, and commercial weight loss programs. Specifically, participants will be asked to report their level of interest in each treatment option on a scale from 1(Not interested) to 5(Very interested).
Ambivalence | 0, 6, 12 months
  All participants will complete the Goal Ambivalence Scale (GAS) (Fadardi et al., 2022) at BL, 6 months, and 12 months. Participants will answer three questions assessing their readiness to lose weight on a scale from 1(Strongly disagree) to 4(Strongly agree). A lower score will indicate more ambivalence, whereas a higher score will indicate less ambivalence and more readiness.
Attitude toward weight management medications | 0, 6, 12 months
  A list of questions developed by Algarni et al. (2023) will be administered to all participants at BL, 6 months, and 12 months. Given the novelty of anti-obesity medications and the controversy surrounding their use and access, these questions will assess participant attitudes towards these medications. Participants will be asked to respond to six statements about weight management medications on a scale from 1(Disagree) to 3(Agree). A score between 8-15 indicates unfavorable attitudes towards weight management medications, while a score >16 indicates favorable attitudes.
Barriers to weight loss medication adherence and uptake | 0, 6, 12 months
  All participants will be administered an adapted version of the Identification of Medication Adherence Barriers Questionnaire (IMAB-Q; Bhattacharya et al., 2023) at BL, 6 months and 12 months. These questions assess participant beliefs about consequences, emotions, and social influences related to medication adherence on a scale from 1(Strongly disagree) to 5(Strongly agree) with 1 indicating that the respondent did not consider the behavioural domain to be a barrier to adherence whilst 5 indicates that it is perceived to be a strong barrier.
MATCH | 0, 6, 12 months
  All participants will complete the Motivation and attitudes towards changing health (MATCH) instrument at BL, 6 months, and 12 months. Participants will respond to statements measuring their willingness, ability, and how worthwhile it is for them to change their weight on a scale from 1(Strongly disagree) to 5(Strongly agree). A higher score indicates that participants are more willing, able, and feel its more worthwhile to change their weight.
Multidimensional trust in healthcare systems | 0, 6, 12 months
  All participants will complete the multidimensional trust in health care systems scale (Egede et al., 2008) at BL, 6 months, and 12 months. Participants will report their level of agreement with statements assessing their trust in health care institutions, health care providers, and health care payers on a scale from 1(Strongly disagree) to 5(Strongly agree). Higher total scores and higher subscale stores represent greater trust in health care systems.
Beliefs and perspectives on obesity | 0, 6, 12 months
  A series of questions developed by Grannell et al. (2021) will be administered to participants at BL, 6 months, and 12 months. These questions will assess participant views on obesity, and participants will be asked to report how much they agree with these statements on a scale from 1(Completely disagree) to 5(Completely agree).
All Aspects of Health Literacy Scale (AAHLS) | 0, 6, 12 months
  All participants will complete the AAHLS, developed by Chinn & McCarthy (2013) at BL, 6 months, and 12 months. These questions assess functional and critical health literacy on a scale from 1(Rarely) to 3(Often). Higher scores indicate greater health literacy.
Weight Loss Self-Efficacy | Baseline, 6 months, 12 months
  Participants will be asked how confident they are in their ability to lose weight in the next 3 months on a scale from 1 (not at all confident) to 10 (very confident). This questions was adapted from Hoeppner et al. (2011)

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel university, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifiable data will be de-identified prior to submission in the public repository to protect research participant privacy and confidentiality. All individual-participant level data will be preserved and shared, as all variables collected are pertinent to scientific questions.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: In accordance with NCI policy, the scientific data will be shared within 12 months of trial completion. Any data included in associated manuscripts will be available at the time of publication; all other scientific data will be shared no later than the end of the award performance period. The study data will be stored in the repository for at least 10 years after the end of the funding period.
Access Criteria: There are no anticipated factors or limitations on access, distribution, or reuse of the scientific data from this proposal. We will address data management and sharing processes during the informed consent process, and all research participants will be consented for broad data sharing of de-identified data.
URL: https://shorturl.at/HzyMB

DOCUMENTS (1):
  • Informed Consent Form (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT06972381/ICF_001.pdf